CLINICAL TRIAL: NCT03476590
Title: A New Model of Medical Care With Use of Modern Methods of Non-invasive Clinical Assessment and Telemedicine in Patients With Heart Failure
Brief Title: New Model of Care in Heart Failure
Acronym: AMULET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Collaborators: Wroclaw Medical University (Other); 4th Military Clinical Hospital with Polyclinic, Poland (Other); Medical University of Gdansk (Other); Military University of Technology (Unknown)
Responsible Party: Principal Investigator, Paweł Krzesiński, Head of Department of Cardiology and Internal Diseases, Military Institute od Medicine National Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STRATEGMED3/305274/8/NCBR/2017
Record Dates: First submitted 2018-03-17; First posted 2018-03-26 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
Keywords: heart failure; ambulatory care; telemedicine; impedance cardiography
MeSH Terms: conditions — Heart Failure | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: prospective, randomized (1:1), open-label and controlled, parallel group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (No Intervention): In standard care group the patients will be recommended to visit physician/cardiologists in standard healthcare system. Two non-interventional visits will be performed: recruitment visit (day of enrolment) and summary visit (12th month after the enrolment)
- intervention group (Experimental): In intervention group patients will be referred to ambulatory care point (ACP) and the physicians will perform remote teleconsultations. The visits will be realized by nurses supported with vital sign assessment based on bioimpedance diagnostic methods (impedance cardiography, bioimpedance scale). The ambulatory visits will be performed according to the schedule: (1') recruitment visit (1st day of enrolment) performed by physician -> 7 ambulatory visits: (1) 1st day of enrolment (performed by nurse and physician), (2) 7th-10th day (performed by nurse and physician), (3) 1st month, (4) 3th month, (5) 6th month, (6) 9th month, (7) 12th month after the enrolment (visits no 3-7 performed by nurse with tele-supervision by physician) and -> (7') summary visit (12th month after the enrolment) performed by physician.
  The plan of visits may be modified if required by the clinical status change, i.e. deterioration of clinical parameters and interim hospitalizations for worsening heart failure.
  Interventions: Procedure: new model of ambulatory care with use of of non-invasive vital signs assessment and telemedicine

INTERVENTIONS:
Procedure: new model of ambulatory care with use of of non-invasive vital signs assessment and telemedicine — The report of symptoms and physical examination will be obligatory performed by the ACP nurse. Self-condition and quality of life assessment at every visit will be based on EQ-5D questionnaire and VAS 10-points scale Hemodynamic assessment - the ACP nurse will perform impedance cardiography (cardiomonitor) and bioimpedance (scale). The parameters measured by ICG and bioimpedance will be assessed with respect to individually defined target values for: heart rate (HR), systolic and diastolic blood pressure (SBP and DBP), thoracic fluid content (TFC) and its change (delta TFC), change of body mass and total body water (delta TBW).
  Supervising physician will confront ICG/bioimpedance results with the patient's clinical data and give final remote recommendations.
  Other Names: Patient's tailored ambulatory care based on remote telemonitoring
  Arms: intervention group

SUMMARY:
Heart failure (HF) is characterized by high mortality, poor quality of life and frequent hospitalizations. The effectiveness of out-patient care for HF patients is unsatisfactory. Therefore the solutions that enable effective monitoring and assessment of HF patients' clinical status become priority in treatment strategy. The applicant proposes to develop a model of care for HF patients based on modern non-invasive diagnostic tools and telemedicine. Clinical evaluation will be based on i.e. impedance cardiography, a simple non-invasive method of hemodynamic monitoring, including assessment of heart rate, blood pressure, left ventricular stroke volume, chest and total fluid status. The telemedicine system will enable rapid, appropriate to the patient's clinical status, therapeutic decision undertaken remotely by specialist. Implementation of the proposed model of care will contribute to a significant improvement in prognosis of HF patients (through i.e. improved access to specialist consultation, the early diagnosis of the deterioration of HF and the optimization of treatment). The significant economic, social and scientific benefits related to the project are also expected.

DETAILED DESCRIPTION:
Treatment of patients with heart failure (HF) is a great challenge for contemporary medicine. HF frequency in European population is assessed for 0.4-2%. This disease is characterized by high morbidity and mortality rate, poor quality of life and frequent hospitalizations. Along with the medicine progress, in particular in the scope of acute coronary syndromes treatment, the number of HF patients is constantly growing. The essential problem connected with HF is its progress course and an increasing rate of subsequent hospitalizations (approximately 30% of hospitalizations are the repeated ones). It is estimated that the costs of hospital stays constitute nearly 2/3 of healthcare costs provided for HF patients.

It has been estimated that the prevalence of HF will increase by 25% and its direct costs by 215% in the next 20 years. The prognosis in HF is closely connected with the progression of the disease defined in accordance with the NYHA (New York Heart Association) functional classification. The yearly mortality rate among each NYHA class is: class 1 - up to 10%, class 2 - 10-20%, class 3 - 20-40%, class 4 - mortality 40-60%. Over a half of the patients with symptomatic HF die within 4 years of observation.

In the AMULET study we we will merging the interventions that so far turned out to be effective (specialist counselling, phone counselling programmes and telemonitoring). Therefore, we created of ambulatory care points for HF patients, which would be equipped with diagnostic devices (impedance cardiography and body composition analyser (bioimpedance scale)), assessing the most important clinical parameters. Ambulatory care point will be operated by a trained nurse, under a telemetry supervision of a specialist.

The following parameters were identified as the indicators of treatment effects: heart rate (HR), systolic and diastolic blood pressure (SBP and DBP), thoracic fluid content (TFC) and its change (delta TFC), change of body mass and total body water (delta TBW).

The telemedicine solutions will strongly support the proposed system. The clinical data will be automatically entered into an interactive system (database), which will send information to a supervising cardiologist, in accordance with the previously implemented recommendation support module (RSM). Regarding RSM indications remote specialist recommendation will be generated (e.g. maintenance or modification of treatment, referral to hospital).

The proposed approach will satisfy ESC recommendations on long-term management: plan follow-up strategy (including plan to up-titrate/optimize dose of disease-modifying drugs); improvement in symptoms, quality of life and survival; prevention of readmissions; management programme; education and appropriate lifestyle adjustments.

ELIGIBILITY:
Inclusion Criteria:

1. age >18 years;
2. HF with LVEF≤49% and at least 1 hospitalization due to the acute HF decompensation (with clinical presentation in NYHA class III-IV) within the last 6 months before enrollment.

Exclusion Criteria:

1. cardiogenic shock
2. myocardial (STE-ACS/NSTE-ACS) infarct as the main cause of hospitalization within the last 40 days prior to recruitment;
3. stroke within 40 days prior to recruitment;
4. cardiac surgery within 90 days prior to recruitment;
5. elective cardiac surgery (or any other high risk surgery) within next 90 days;
6. pulmonary embolism within 40 days prior to recruitment;
7. severe pulmonary diseases, including: chronic obstructive pulmonary disease (stage C/D), uncontrolled asthma, pulmonary hypertension (WHO class III-IV);
8. chronic kidney disease (stage 5 and/or requiring dialysis);
9. severe inflammatory disease, including: pneumonia as the main cause of hospitalization; sepsis; tuberculosis;
10. severe mental and physical disorders;
11. life expectancy less than 12 months in the opinion of the physician because of reasons other than HF;
12. patient currently enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study (ies), or subject is receiving other investigational agent(s).
13. pregnancy;
14. patients' refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
cardiovascular death and/or hospitalization for worsening heart failure (HF). | 12 months

SECONDARY OUTCOMES:
cardiovascular death | 12 months
death due to worsening of HF | 12 months
all-cause death | 12 months
hospitalization for worsening HF | 12 months
cardiovascular hospitalization | 12 months
all-cause hospitalization | 12 months
number of hospitalizations for worsening HF per patient during 12 months of follow-up | 12 months
days lost due to unplanned HF hospitalisation(s) or all-cause mortality | 12 months

OTHER OUTCOMES:
time to first hospitalization for any reason | 12 months
time to first hospitalization for any cardiovascular reason | 12 months
time to first hospitalization due to worsening HF | 12 months
time to death for any reason | 12 months
time to death for any cardiovascular reason | 12 months
time to death due to worsening HF | 12 months
SF-36 score at 12 months adjusted for baseline | 12 months
Minnesota Questionnaire score at 12 months adjusted for baseline | 12 months
NYHA functional class at 12 months adjusted for baseline | 12 months
final (12 month) daily doses (% of guidelines required target dose) of the following medicaments: ACEI, ARB, beta-blocker, MRA, ARNI | 12 months
final (12 month) doses (mg) of the diuretics (furosemide, torasemide, hydrochlorotiazide, indapamid) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Military Institute of Medicine, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krzesinski P, Siebert J, Jankowska EA, Banasiak W, Piotrowicz K, Stanczyk A, Galas A, Walczak A, Murawski P, Chrom P, Gutknecht P, Siwolowski P, Ponikowski P, Gielerak G. Rationale and design of the AMULET study: A new Model of telemedical care in patients with heart failure. ESC Heart Fail. 2021 Aug;8(4):2569-2579. doi: 10.1002/ehf2.13330. Epub 2021 Apr 22. PMID 33887120